CLINICAL TRIAL: NCT06230731
Title: Oxygenation in Vascular Lesions of the Colon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB23-1273
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Vascular Lesion
MeSH Terms: interventions — Oxygen Saturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vascular abnormality group (Experimental): People with acquired vascular abnormalities in the proximal colon
  Interventions: Other: Oxygen saturation
- Control group (Active Comparator): People with healthy colon
  Interventions: Other: Oxygen saturation

INTERVENTIONS:
Other: Oxygen saturation — Measure oxygen levels in 5 proximal colon mucosa locations.

SUMMARY:
The goal of this clinical trial is to evaluate oxygenation in the colon in people with acquired vascular abnormalities in the proximal colon.

DETAILED DESCRIPTION:
The etiology of acquired vascular abnormalities of the large bowel (i.e. angiodysplasia, AVM, hemangiomas of the cecum. etc.) are unknown. These lesions typical appear as ectatic, dilated, and tortuous blood vessels within the submucosa and mucosa of the GI tract. In some patients they are the cause of acute large volume bleeding or a slower chronic bleed that manifests as chronic iron deficiency anemia. These lesions are more common in older individuals and those with underlying cardiac, pulmonary, and renal disease. As such, it is hypothesized that these lesions may result from chronic hypoxia. This study aims to evaluate oxygenation of the colon in people with acquired vascular abnormalities in the proximal colon compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Undergo standard of care colonoscopy
* People with a history of vascular lesions of the colon
* People with healthy colon
* 18 - 89 years of age

Exclusion Criteria:

* Age < 18 years
* Age > 90 years
* People with ulcerations in at ascending colon opposite the ileocecal valve
* Previous colon surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis of colonic oxygen saturation levels | baseline-12 months
  Colonic oxygen saturation levels will be compared between patients with vascular lesions of the colon and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Pekow, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No